CLINICAL TRIAL: NCT05083455
Title: Replication of the RECORD1 Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-RECORD1
Record Dates: First submitted 2021-09-20; First posted 2021-10-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Deep Vein Thrombosis, Pulmonary Embolus
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Enoxaparin: Reference group
  Interventions: Drug: Enoxaparin
- Rivaroxaban: Exposure group
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Any rivaroxaban dispensing claim is used as the exposure group
  Other Names: Xarelto
  Groups: Rivaroxaban
Drug: Enoxaparin — Any enoxaparin dispensing claim is used as the reference group
  Groups: Enoxaparin

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates through standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Inclusion Criteria:

* At least 18 years of age
* Scheduled to undergo elective total hip arthroplasty

Exclusion Criteria:

* Scheduled to undergo staged, bilateral hip arthroplasty [Day -30, Day 0]
* Pregnany or breastfeeding [Day -180, Day 0]
* Had active bleeding or high risk of bleeding [Day -180, Day 0]
* Had conditions preventing bilateral venography [Day -30, Day 0]
* Congestive heart failure [Day -180, Day 0]
* Pulmonary hypertension [Day -180, Day 0]
* Edema of legs [Day -180, Day 0]
* Substantial liver disease [Day -180, Day 0]
* Severe renal impairment (creatinine clearance <30 ml per minute) [Day -180, Day 0]
* Concomitant use of protease inhibitors for the treatment of HIV [Day -180, Day 0]

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing rivaroxaban to enoxaparin users. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of rivaroxaban or enoxaparin (index date). We will restrict the analyses to patients who underwent a total hip arthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 89215 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Relative hazard of any deep vein thrombosis, non-fatal pulmonary embolism, or death from any cause | Through study completion or censoring, up to 36 days
  Claims-based algorithm: relative hazard of any deep vein thrombosis, non-fatal pulmonary embolism, or death from any cause.

SECONDARY OUTCOMES:
Relative hazard of major bleeding | Through study completion or censoring, up to 36 days
  Claims-based algorithm: relative hazard of major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT05083455/Prot_000.pdf